CLINICAL TRIAL: NCT03143556
Title: Comparison of Cystoscopic Removal Versus Magnetic Device Removal of Ureteral Stents in Renal Transplant Recipients
Brief Title: Black Star - Magnetic Stent Removal in Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Anil Kapoor, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07282016
Record Dates: First submitted 2017-04-05; First posted 2017-05-08 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2019-05

CONDITIONS: Kidney Failure, Chronic; End Stage Renal Failure With Renal Transplant
Keywords: renal transplant; magnetic ureteral stent; Black-Star®
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic Stent (Experimental): Patients who are undergoing renal transplant surgery for the treatment of end stage renal failure and randomized for magnetic stent group will receive magnetic stent and the removal of stent would be done by help of magnetic device.
  Interventions: Device: Magnetic stent
- Routine stent (No Intervention): Patients who are undergoing renal transplant surgery for the treatment of end stage renal failure and randomized for routine stent would receive routine stent and the removal of stent would be done by cystoscopy

INTERVENTIONS:
Device: Magnetic stent — Patients who are undergoing renal transplant surgery for the treatment of end stage renal failure will be assigned to magnetic stent or routine stent using computer generated randomization method in the operating room. Those who receive magnetic stent would get their stent removal by magnetic device retrieval and not by routine cystoscopy.
  Other Names: Black-Star®
  Arms: Magnetic Stent

SUMMARY:
This is a pilot, single-centre, feasibility study to assess the feasibility issues and collect preliminary clinical data for the design of future randomized controlled trial to evaluate the feasibility and patient comfort of magnetic retrieval device removal of ureteral stent in transplant patients.

DETAILED DESCRIPTION:
To curtail the pain and discomfort during cystoscopic stent removal and in order to improve patient's quality of life, a newly developed ureteral stent with a small magnet at its distal end and a customized magnetic retrieval catheter is recently used in Europe. The product is Black-Star® with a retrieval device by Urotech (Achenmühle, Germany). The magnetic Blackstar stent is a ureteral stent with a small magnet fixed with a string at the distal loop. The placement of stent is similar as routinely done on a guidewire, the only difference is to include the magnetic piece over the guidewire. To remove the stent a customized catheter with a magnetic Tiemann tip is used. The catheter is inserted after urethral application of a standard lubricant and removed with the stent after coming in contact with the stent's magnet.

The stent comes in various sizes and is currently being used in Europe. The studies have concluded fast and easy retrieval of stent without requirement of cystoscopy and decreased patient discomfort.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years of age and capable of giving informed consent
2. Patients scheduled for deceased donor renal transplant surgery

Exclusion Criteria:

1) Patients undergoing Live donor renal transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Feasibility and patient comfort of the retrieval device, using standard validated questionnaire Ureteral Stent Symptom Questionnaire (USSQ) | 3-6 weeks
  All patients will be followed up 4 weeks post renal transplant surgery, until ureteral stent removal. Feasibility and comfort of stent retrieval, Ureteral Stent Symptom Questionnaire (USSQ) at 4 weeks before stent removal and 1 week post stent removal.

SECONDARY OUTCOMES:
Outcome measure: Retrieval time | Baseline (intraoperatively)
  Retrieval time in minutes: The time taken for ureteric stent removal (both routine and magnetic stent) will be documented and mean time taken will be calculated. This will show which technique takes less time.
Outcome measure: Infection rate | 3-6 weeks
  Infection rates: Number of Urine culture positive with stent in situ and after removal of stent (both routine and magnetic stent). This will suggest if magnetic stent is associated with an increased incidence of urinary tract infections as compared to the routine stent.
Outcome measure: Cost effectiveness | 3-6 weeks
  Cost effective analysis: Units will be Canadian Dollars; we will analyze the cost of disposables, sterilization of instruments, use of cystoscopy suite and also nursing and surgeon charges. Mean cost taken for either procedure will be compared to find cost effectiveness

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Theckumparampil N, Elsamra SE, Carons A, Salami SS, Leavitt D, Kavoussi A, Motola J, Smith A, Okeke Z. Symptoms after removal of ureteral stents. J Endourol. 2015 Feb;29(2):246-52. doi: 10.1089/end.2014.0432. Epub 2014 Sep 17. PMID 25137344
- [Background] Kumar A, Kumar R, Bhandari M. Significance of routine JJ stenting in living related renal transplantation: a prospective randomised study. Transplant Proc. 1998 Nov;30(7):2995-7. doi: 10.1016/s0041-1345(98)00902-6. No abstract available. PMID 9838320
- [Background] Wilson CH, Bhatti AA, Rix DA, Manas DM. Routine intraoperative stenting for renal transplant recipients. Transplantation. 2005 Oct 15;80(7):877-82. doi: 10.1097/01.tp.0000181197.21706.fa. PMID 16249733
- [Background] Englesbe MJ, Dubay DA, Gillespie BW, Moyer AS, Pelletier SJ, Sung RS, Magee JC, Punch JD, Campbell DA Jr, Merion RM. Risk factors for urinary complications after renal transplantation. Am J Transplant. 2007 Jun;7(6):1536-41. doi: 10.1111/j.1600-6143.2007.01790.x. Epub 2007 Apr 8. PMID 17430402
- [Result] Mangus RS, Haag BW. Stented versus nonstented extravesical ureteroneocystostomy in renal transplantation: a metaanalysis. Am J Transplant. 2004 Nov;4(11):1889-96. doi: 10.1111/j.1600-6143.2004.00595.x. PMID 15476491